CLINICAL TRIAL: NCT03120130
Title: Phase I Study (First in Humans) of the Amblyomin-X in the Treatment of Patients With Advanced Solid Tumors Refractory or Without Indication / Access to Standard Treatment
Brief Title: Study of Amblyomin-X in Advanced Solid Tumor
Acronym: Amblyomin-X
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Delay in the R & D stage
Sponsor: União Química Farmacêutica Nacional S/A (Industry)
Collaborators: Buranello e Rodrigues Consultoria em Desenvolvimento Farmacêutico Ltda ME (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PGUQ002
Record Dates: First submitted 2017-03-29; First posted 2017-04-19 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-06

CONDITIONS: Advanced Cancer
Keywords: Phase I,
MeSH Terms: interventions — Amblyomin-X protein, Amblyomma cajennense

STUDY DESIGN:
Intervention Model Description: Study with dose escalation regime, done according to the classic scheme known as "3 + 3"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): This cohort will include 3 patients with the first calculated dose of Amblyomin-X drug. The patient will receive the intravenous drug. If no Dose-limiting toxicity (DLT) in this group the study continues including the next cohort. However, if If only one patient in a given cohort develops DLT, three more patients will be included at that dose level, up to a maximum total of six patients per dose level. If two or more of the three patients of a certain dose level develop DLT, this dose level is considered very toxic, and the study does not proceed. If this occurs at the first dose level, the study will be finalized. If only one in six patients at a dose level develops DLTs, escalation proceeds until Tolerated Maximum Dose.
  Interventions: Biological: Amblyomin-X
- Cohort 2 (Experimental): This cohort will include 3 patients with the second calculated dose of Amblyomin-X drug. The patient will receive the intravenous drug. If no Dose-limiting toxicity in this group the study continues including the next cohort
  Interventions: Biological: Amblyomin-X
- Cohort 3 (Experimental): This cohort will include 3 patients with the third calculated dose of Amblyomin-X drug. The patient will receive the intravenous drug. If no Dose-limiting toxicity in this group the study continues including the next cohort
  Interventions: Biological: Amblyomin-X
- Cohort 4 (Experimental): This cohort will include 3 patients with the fourth calculated dose of Amblyomin-X drug. The patient will receive the intravenous drug. If no Dose-limiting toxicity in this group the study continues including the next cohort
  Interventions: Biological: Amblyomin-X
- Cohort 5 (Experimental): This cohort will include 3 patients with the fifth calculated dose of Amblyomin-X drug. The patient will receive the intravenous drug. If no Dose-limiting toxicity in this group the study continues including the next cohort
  Interventions: Biological: Amblyomin-X
- Cohort 6 (Experimental): This cohort will include 3 patients with the sixth calculated dose of Amblyomin-X drug, the last dose calculated. The patient will receive the intravenous drug.
  Interventions: Biological: Amblyomin-X

INTERVENTIONS:
Biological: Amblyomin-X — Intravenous drug administration, with different doses in each cohort

SUMMARY:
Amblyomin-X is an inhibitor of Factor Xa that also acts as an apoptotic agent for tumor cells. In the case of in vitro assays, Amblyomin-X induces tumor cells to death and does not affect the viability of normal cells. When in vivo assays were performed on mice bearing tumors, treatment with Amblyomin-X caused a significant reduction in tumor mass and number of metastases.

DETAILED DESCRIPTION:
This trial will be the first clinical study in humans with the product, which until then has been studied only in experimental models. Given the current epidemiological impact of cancer and the need to improve its systemic treatment, making it available to a larger portion of the Brazilian population, it is proposed to conduct the first Amblyomin-X study in cancer patients, more specifically those with advanced solid tumors For which there is no contraindicated or inaccessible therapeutic option established as the standard at the time of inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must sign the Free and Informed Consent Term (TCLE),
* be between 18 and 75 years of age,
* present a solid tumor proven by anatomopathological examination at an advanced or metastatic stage and refractory to conventional treatment or without current indication or access to conventional treatment ,
* have a life expectancy of at least 12 weeks.
* presence of measurable disease according to Response Response Criteria in Solid Tumors (RECIST, version 1.1),
* medullary, renal and hepatic functions within acceptable limits (defined in protocol),
* end of the previous antineoplastic treatment at least 4 weeks (since the last dose of any antineoplastic medication, radiotherapy, or surgical procedure).

Exclusion Criteria:

* The presence of previously non-irradiated brain metastasis;
* Prediction of the use of radiotherapy, surgery, systemic antineoplastic treatment, or any other form of treatment for cancer after inclusion in the study;
* Prediction of corticosteroid use, hematopoietic growth factors or inhibitors of bone resorption during the first course of treatment (4 weeks);
* Regular use of anticoagulants or known previous coagulation disorder;
* Severe comorbidity (at the discretion of the researcher);
* Gestational, lactating, pregnant women, or who have not been surgically infertile or menopausal for at least 12 months;
* Men and women who refuse to use an adequate contraceptive method during the study period;
* Participation of another clinical study in the last 12 months (unless justified by the investigator);
* Or inability to comply with study requirements and procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-08-20 (Estimated); Study Completion 2022-05-22 (Estimated)

PRIMARY OUTCOMES:
grade 4 or non-haematological grade 3 haematological toxicity according to the CTCAE (version 4) | 2 weeks
  Presence of grade 4 or non-haematological grade 3 haematological toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4)

SECONDARY OUTCOMES:
maximum tolerated dose (MTD) and the recommended dose for phase II | 2 weeks
  This will be based on dose-limiting toxicity of the previous cohort
Adverse Events | 4 weeks
  haematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Paula F Santos, Study Director — União Quimica
Locations (1):
- União Química Farmacêutica Nacional, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No